CLINICAL TRIAL: NCT05336331
Title: Establishing Laparoscopic Sleeve Gastrectomy as a Standard Procedure at a Swedish Bariatric Center
Brief Title: Sleeve Gastrectomy as a Standard Bariatric Procedure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: YCengiz
Record Dates: First submitted 2022-02-14; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Complications
Keywords: bariatric surgery; laparoscopic Roux-en-Y gastric bypass; laparoscopic sleeve gastrectomy; Morbid obesity; Weight loss; Metabolic control; Metabolic syndrome; Complication risk
MeSH Terms: conditions — Postoperative Complications; Obesity, Morbid; Weight Loss; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic sleeve gastrectomy (SG): Patients operated on with a SG
  Interventions: Procedure: SG or a RYGB
- laparoscopic Roux-en-Y gastric bypass (RYGB): patients operated on with aRYGB
  Interventions: Procedure: SG or a RYGB

INTERVENTIONS:
Procedure: SG or a RYGB — operation type differed between a partial gastrectomy (SG)or a combined restrictive/malabsorptive

SUMMARY:
This study compared differences in weight loss, comorbidity resolution and complications and reoperations between a recently established sleeve gastrectomy (SG) and prior laparoscopic Rox-en-Y gastric bypass (RYGB).

DETAILED DESCRIPTION:
This retrospective study with prospectively collected registry data presents results from establishment of SG as standard procedure for morbid obesity. Our first 368 patients operated with a SG were compared to 647 patients previously operated with a (RYGB. Perioperative data and results up to 2 years postoperatively regarding weight control, metabolic control as well as complications/reoperations necessary were registered.

In summary, a RYGB was associated with a longer operation time and higher rates of late complications and reoperations. Diabetes resolution was similar in both groups but patients with a RYGB had greater weight loss and significant improvement in hypertension and dyslipidemias.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either a BMI 35 or higher with comorbidity, or patients with a BMI of 40 or more without known comorbidity associated, undergoing a primary laparoscopic bariatric surgery in Sundsvall,Sweden 2010-01-01 to 2018-06-10.

Exclusion Criteria:

* All other patients undergoing a bariatric surgery during this time frame

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Morbid obesity patients found suitable for a SG or RYGB
Sampling Method: Non-Probability Sample
Enrollment: 1015 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss | after 6 weeks
  weight and height will be combined to report various measurements of BMI in kg/m^2
Weight loss | after 1 year
  weight and height will be combined to report various measurements of BMI in kg/m^2
Weight loss | after 2 years
  weight and height will be combined to report various measurements of BMI in kg/m^2
Changes in Diabetes | after 1 year
  measured as fasting plasma glucose and/or Hemoglobin A1c
Changes in Diabetes | after 2 years
  measured as fasting plasma glucose and/or Hemoglobin A1c
Changes in Hypertension | after 1 year
  measured as Systolic- and Diastolic Blood Pressure
Changes in Hypertension | after 2 years
  measured as Systolic- and Diastolic Blood Pressure
Changes in hypertriglyceridemia (plasma-level >1.7 mmol/l) | after 1 year
  measured as hypertriglyceridaemia (plasma-level >1.7 mmol/l)
Changes in hypertriglyceridemia (plasma-level >1.7 mmol/l) | after 2 year
  measured as hypertriglyceridaemia (plasma-level >1.7 mmol/l)
Changes in Hypercholesterolemia (LDL-C > 3.0 mmol/L and/or HDL-C < 1.0 mmol/L). | after 1 years
  Measured as Hypercholesterolemia (Plasma concentration of LDL >3.0 mmol/L and/or of HDL < 1.0 mmol/L).
Changes in Hypercholesterolemia (LDL-C > 3.0 mmol/L and/or HDL-C < 1.0 mmol/L). | after 2 years
  Measured as Hypercholesterolemia (Plasma concentration of LDL >3.0 mmol/L and/or of HDL < 1.0 mmol/L).
Duration of surgery | From the start of the operation until completion, in average 62 minutes
  Operation time in minutes
Duration of hospital stay | From time of operation until discharge, in average 1.7 days
  Duration of hospital stay in days
Early complications | At six weeks
  Complications occurred until six weeks from operation
Early reoperations | At six weeks
  Reoperations occurred until six weeks from operation
Late complications | From six weeks until 2 years from operation
  Complications occurred from six weeks until 2 years from operation
Late reoperations | From six weeks until 2 years from operation
  Reoperations occurred from six weeks until 2 years from operation

CONTACTS AND LOCATIONS:
Locations (1):
- Sundsvall Hospital, Sundsvall, Sweden

IPD SHARING:
Plan to Share IPD: No